CLINICAL TRIAL: NCT07300891
Title: T Cell Inflamed Gene Expression Profiling Score-guided Anti PD-1 Therapy (Tislelizumab Monotherapy) for Refractory Solid Cancer Patients Unexposed to Immunotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Se-Hoon Lee, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAN-IO-001
Record Dates: First submitted 2025-12-02; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Refractory Solid Cancer Patients Unexposed to Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab(BGB-A317) (Experimental)
  Interventions: Drug: Tisleizumab(BGB-A317)

INTERVENTIONS:
Drug: Tisleizumab(BGB-A317) — T cell inflamed GEP score

SUMMARY:
This is a Phase 2, single-arm, multicenter study, evaluating the anti-tumor efficacy of tumor-infiltrating lymphocyte (TIL) directed tislelizumab monotherapy (also known as BGB-A317) for refractory solid tumors in approximately 72 patients with centrally confirmed T cell inflamed GEP score ≥ 0.857, who have not been previously exposed to immunotherapy.

All patients must provide a tumor specimen for T cell inflamed GEP assessment. Archived tissue slide collected within 2 years from the first dose of study drug must be provided.

This study will include a Screening Period, a Treatment Period, and a Follow-Up Period. All patients will complete up to 28 days of screening. During the Treatment Period, patients will receive tislelizumab 200 mg fixed dose once every 3 weeks by intravenous (IV) administration until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.

After treatment discontinuation, patients will be follow-up for disease progression and survival status until death, withdrawal of consent, or study closure, whichever occurs first.

The end of study will be the timepoint when the final data for the study were collected. Additionally, the Investigator Sponsor has the right to terminate this study at any time.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 20 years at the time of informed consent.
2. Patients with histologically- or cytologically confirmed advanced or metastatic solid tumor who are no longer benefiting from standard anti-cancer treatment or for whom, in the opinion of site physicians, no such treatment is available or indicated according to local or international guidelines.
3. Centrally confirmed T cell inflamed GEP score ≥ 0.857 assessed by RNA sequencing. For baseline T cell inflamed GEP, an archived tissue sample collected within 2 years from the first dose of study drug must be provided. T cell inflamed gene expression profiling will be assessed at a central laboratory. Patients who have at least 1 target lesion per the Response Evaluation Criteria in Solid Tumors (RECIST) Guideline Ver. 1.1 as confirmed by imaging within 28 days before first dose of study drug.
4. ECOG Performance Status Score 0 or 1.
5. Patients with a life expectancy of at least 3 months.
6. Patients with adequate hematological and biological function as indicated by the following screening laboratory values:

   * Absolute neutrophil count (ANC) ≥ 1.5×109/L
   * Platelets ≥ 75×109/L
   * Hemoglobin ≥ 9g/dL or ≥ 5.6 mmol/L (Note: Criteria must be met without a transfusion within 14 days of obtaining the sample)
   * Calculated creatinine clearance ≤ 1.5×upper limit of normal (ULN), or estimated GFR ≥ 60 mL/min by Cockcroft-Gault formula
   * Serum total bilirubin ≤ 1.5×ULN (total bilirubin must be < 3×ULN for patients with Gilbert's syndrome)
   * Aspartate aminotransferase (AST) and ALT ≤ 3×ULN OR ≤ 5×ULN for patients with liver metastases

Exclusion Criteria:

1. Patients aged ≥ 20 years at the time of informed consent.
2. Patients with histologically- or cytologically confirmed advanced or metastatic solid tumor who are no longer benefiting from standard anti-cancer treatment or for whom, in the opinion of site physicians, no such treatment is available or indicated according to local or international guidelines.
3. Centrally confirmed T cell inflamed GEP score ≥ 0.857 assessed by RNA sequencing. For baseline T cell inflamed GEP, an archived tissue sample collected within 2 years from the first dose of study drug must be provided. T cell inflamed gene expression profiling will be assessed at a central laboratory. Patients who have at least 1 target lesion per the Response Evaluation Criteria in Solid Tumors (RECIST) Guideline Ver. 1.1 as confirmed by imaging within 28 days before first dose of study drug.
4. ECOG Performance Status Score 0 or 1.
5. Patients with a life expectancy of at least 3 months.
6. Patients with adequate hematological and biological function as indicated by the following screening laboratory values:

   * Absolute neutrophil count (ANC) ≥ 1.5×109/L
   * Platelets ≥ 75×109/L
   * Hemoglobin ≥ 9g/dL or ≥ 5.6 mmol/L (Note: Criteria must be met without a transfusion within 14 days of obtaining the sample)
   * Calculated creatinine clearance ≤ 1.5×upper limit of normal (ULN), or estimated GFR ≥ 60 mL/min by Cockcroft-Gault formula
   * Serum total bilirubin ≤ 1.5×ULN (total bilirubin must be < 3×ULN for patients with Gilbert's syndrome)
   * Aspartate aminotransferase (AST) and ALT ≤ 3×ULN OR ≤ 5×ULN for patients with liver metastases

Key exclusion criteria Patients who meet any of the following criteria at the time of assessment will be excluded.

1. Patients with solid tumors from multiple primary origin (with the exception of completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, or superficial bladder cancer, or any other cancer that has not recurred for at least 3 years).
2. Patients with residual adverse effects of prior therapy or effects of surgery that would affect the safety evaluation of the investigational product in the opinion of the investigator or sub-investigator.
3. Patients are expected to require any other form of systemic or localized antineoplastic therapy while on trial (including radiation therapy, and/or surgical resection).
4. Patients who have previously received treatment with PD-1/PD-L1 inhibitor or CTLA-4 inhibitor e.g. pembrolizumab, nivolumab, cemiplimab, atezolizumab, avelumab, durvalumab, tislelizumab, dostarlimab, spartalizumab tremelimumab or ipilimumab
5. Active leptomeningeal disease or uncontrolled brain metastasis. Patients with equivocal findings or with confirmed brain metastases are eligible for enrollment provided that they are asymptomatic and radiologically stable without the need for corticosteroid treatment for ≥ 4 weeks before first dose of study drug.
6. Patients have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study in terms of efficacy and safety, interfere with the subject's participation for the full duration of the trial, or are not in the best interest of the subject to participate, in the opinion of the treating investigator.
7. Women who are pregnant or breastfeeding, or possibly pregnant.
8. Patients who have received any other unapproved drug (e.g., investigational use of drugs, unapproved combined formulations, or unapproved dosage forms) within 28 days before first dose of study drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
ORR in refractory solid tumor patients with T cell inflamed GEP score ≥ 0.857 treated with Tislelizumab | From enrollment to the end of treatment at 30days(+/-7)
  ORR is defined as the proportion of patients who had complete response (CR) or partial response (PR) assessed by investigator using RECIST v1.1

SECONDARY OUTCOMES:
ORR in refractory solid tumor patients with T cell inflamed GEP score ≥ 0.955 treated with Tislelizumab. | From enrollment to the end of treatment at 30days(+/-7)
ORR in refractory solid tumor patients with T cell inflamed GEP score ≥ 1.058 treated with Tislelizumab. | From enrollment to the end of treatment at 30days(+/-7)
OS in refractory solid tumor patients with T cell inflamed GEP score ≥ 0.857 treated with Tislelizumab. | From enrollment to the end of treatment at 30days(+/-7)
  - OS is defined as the time from first dose of study drug until death from any cause.
PFS in refractory solid tumor patients with T cell inflamed GEP score ≥ 0.857treated with Tislelizumab. | From enrollment to the end of treatment at 30days(+/-7)
  PFS is defined as the time from first dose
CBR in refractory solid tumor patients with T cell inflamed GEP score ≥ 0.857treated with Tislelizumab. | From enrollment to the end of treatment at 30days(+/-7)
  CBR is defined as the proportion of patients with best overall response of CR and PR, or at least six months of stable disease, per RECIST v1.1.
DOR in refractory solid tumor patients with T cell inflamed GEP score ≥ 0.857treated with Tislelizumab. | From enrollment to the end of treatment at 30days(+/-7)
  DOR is defined as the time from the first determination of an objective response per RECIST v1.1, until objective tumor progression or death from any cause, whichever occurs first.
iORR in refractory solid tumor patients with T cell inflamed GEP score ≥ 0.857 treated with Tislelizumab. | From enrollment to the end of treatment at 30days(+/-7)
  iORR is defined as the proportion of patients who had CR or PR assessed by investigator using iRECIST
iPFS in refractory solid tumor patients with T cell inflamed GEP score ≥ 0.857 treated with Tislelizumab. | From enrollment to the end of treatment at 30days(+/-7)
  iPFS is defined as the time from first dose of study drug until objective tumor progression per iRECIST or death from any cause, whichever occurs first.
iCBR in refractory solid tumor patients with T cell inflamed GEP score ≥ 0.857 treated with Tislelizumab. | From enrollment to the end of treatment at 30days(+/-7)
  iCBR is defined as the proportion of patients with best overall response of CR and PR, or at least six months of stable disease, per iRECIST.
iDOR in refractory solid tumor patients with T cell inflamed GEP score ≥ 0.857 treated with Tislelizumab. | From enrollment to the end of treatment at 30days(+/-7)
  iDOR is defined as the time from the first determination of an objective response per iRECIST, until objective tumor progression or death from any cause, whichever occurs first.
The safety of Tislelizumab in refractory solid tumor patients per NCI CTCAE v5.0 | From enrollment to the end of treatment at 30days(+/-7)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. However, study results and summary data will be made available through the ClinicalTrials.gov results module and/or peer-reviewed publications.